CLINICAL TRIAL: NCT00441558
Title: Worldwide One-year Open-label Safety Study of Flibanserin in Women With HSDD
Brief Title: A One-year Safety Study of Flibanserin to Treat Pre-Menopausal Women With Hypoactive Sexual Desire Disorder (HSDD).
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated for administrative reasons
Sponsor: Sprout Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 511.84
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2014-06-13 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-05

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — flibanserin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- flibanserin (Experimental): flexible dosing of either 50 or 100mg every evening, or 25 or 50mg twice daily.
  Interventions: Drug: Flibanserin

INTERVENTIONS:
Drug: Flibanserin — flexible dosing of either 50 or 100mg every evening, or 25 or 50mg twice daily.

SUMMARY:
To determine if long-term treatment with Flibanserin is safe and to monitor the effectiveness of Flibanserin in Women with HSDD that have already completed a previous study (511.70/71/.74/.75/.105) with Flibanserin.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a primary diagnosis of HSDD who have completed a previous study of Flibanserin.
2. Patients must have used a medically acceptable method of contraception for at least 2 months before the start of the study and continue to use that method for the duration of the study.
3. Patients must be reliable, compliant, and agree to cooperate with all study evaluations.
4. Patients must be able and willing to give meaningful, written informed consent prior to the start of the study and be willing to discuss their sexual functioning with the study staff.

Exclusion Criteria:

1. A history of Major Depressive Disorder within 6 months prior to the start of the study, current suicidal thoughts, or any history of a suicide attempt.
2. Participation in another clinical trial within 1 month prior to the start of the study, except for Flibanserin.
3. Patients with pelvic inflammatory disease, urinary tract infection, vaginal infection/vaginitis, cervicitis, interstitial cystitis, vulvodynia, or significant vaginal atrophy.
4. Patients who are pregnant or have been pregnant within 1 month prior to study start.
5. Patients experiencing major life stress (including loss of income, death of a family member, major illness, etc.) or relationship trouble that could interfere with sexual activity, except distress about HSDD.
6. Clinically significant ECG or lab abnormalities at study start.
7. Patients taking prohibited medications that were excluded in their previous trial which contribute to sexual dysfunction or safety-related interactions.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1723 (Actual)
Dates: Start 2007-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (196):
- United States (173):
  - 511.84.01079 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.84.01193 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 511.84.01188 Boehringer Ingelheim Investigational Site, Huntsville, Alabama
  - 511.84.01110 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.84.01142 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.84.01157 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 511.84.01162 Boehringer Ingelheim Investigational Site, Little Rock, Alaska
  - 511.84.01070 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.84.01191 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 511.84.01115 Boehringer Ingelheim Investigational Site, Tucson, Arizona
  - 511.84.01013 Boehringer Ingelheim Investigational Site, Jonesboro, Arkansas
  - 511.84.01087 Boehringer Ingelheim Investigational Site, Berkeley, California
  - 511.84.01077 Boehringer Ingelheim Investigational Site, Encinitas, California
  - 511.84.01074 Boehringer Ingelheim Investigational Site, Fair Oaks, California
  - 511.84.01104 Boehringer Ingelheim Investigational Site, Irvine, California
  - 511.84.01037 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 511.84.01056 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 511.84.01195 Boehringer Ingelheim Investigational Site, Sacramento, California
  - 511.84.01043 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.84.01047 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.84.01096 Boehringer Ingelheim Investigational Site, San Diego, California
  - 511.84.01040 Boehringer Ingelheim Investigational Site, Stanford, California
  - 511.84.01048 Boehringer Ingelheim Investigational Site, Tarzana, California
  - 511.84.01017 Boehringer Ingelheim Investigational Site, Torrance, California
  - 511.84.01173 Boehringer Ingelheim Investigational Site, Vista, California
  - 511.84.01029 Boehringer Ingelheim Investigational Site, Walnut Creek, California
  - 511.84.01137 Boehringer Ingelheim Investigational Site, Westlake Village, California
  - 511.84.01090 Boehringer Ingelheim Investigational Site, Aurora, Colorado
  - 511.84.01164 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.84.01184 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 511.84.01004 Boehringer Ingelheim Investigational Site, Englewood, Colorado
  - 511.84.01006 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 511.84.01138 Boehringer Ingelheim Investigational Site, Farmington, Connecticut
  - 511.84.01044 Boehringer Ingelheim Investigational Site, Groton, Connecticut
  - 511.84.01016 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 511.84.01108 Boehringer Ingelheim Investigational Site, New Britain, Connecticut
  - 511.84.01168 Boehringer Ingelheim Investigational Site, New London, Connecticut
  - 511.84.01166 Boehringer Ingelheim Investigational Site, Newark, Delaware
  - 511.84.01160 Boehringer Ingelheim Investigational Site, Washington D.C., District of Columbia
  - 511.84.01065 Boehringer Ingelheim Investigational Site, Aventura, Florida
  - 511.84.01005 Boehringer Ingelheim Investigational Site, Boynton Beach, Florida
  - 511.84.01146 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 511.84.01144 Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - 511.84.01169 Boehringer Ingelheim Investigational Site, Daytona Beach, Florida
  - 511.84.01085 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 511.84.01194 Boehringer Ingelheim Investigational Site, Fort Meyers, Florida
  - 511.84.01002 Boehringer Ingelheim Investigational Site, Gainesville, Florida
  - 511.84.01069 Boehringer Ingelheim Investigational Site, Gainsville, Florida
  - 511.84.01007 Boehringer Ingelheim Investigational Site, Hudson, Florida
  - 511.84.01055 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.84.01064 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 511.84.01182 Boehringer Ingelheim Investigational Site, New Port Richey, Florida
  - 511.84.01167 Boehringer Ingelheim Investigational Site, Ocala, Florida
  - 511.84.01111 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.84.01118 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 511.84.01135 Boehringer Ingelheim Investigational Site, Pembroke Pines, Florida
  - 511.84.01032 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 511.84.01175 Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - 511.84.01053 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.84.01132 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 511.84.01117 Boehringer Ingelheim Investigational Site, Stuart, Florida
  - 511.84.01159 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.84.01170 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.84.01183 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 511.84.01003 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.84.01022 Boehringer Ingelheim Investigational Site, West Palm Beach, Florida
  - 511.84.01024 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.84.01061 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.84.01205 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 511.84.01176 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 511.84.01139 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 511.84.01023 Boehringer Ingelheim Investigational Site, Sandy Springs, Georgia
  - 511.84.01179 Boehringer Ingelheim Investigational Site, Champaign, Illinois
  - 511.84.01113 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.84.01165 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.84.01172 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 511.84.01143 Boehringer Ingelheim Investigational Site, Evansville, Indiana
  - 511.84.01092 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 511.84.01202 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 511.84.01049 Boehringer Ingelheim Investigational Site, Lexington, Kentucky
  - 511.84.01025 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 511.84.01171 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 511.84.01192 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 511.84.01130 Boehringer Ingelheim Investigational Site, New Orlean, Louisiana
  - 511.84.01001 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 511.84.01120 Boehringer Ingelheim Investigational Site, Brighton, Massachusetts
  - 511.84.01030 Boehringer Ingelheim Investigational Site, Haverhill, Massachusetts
  - 511.84.01127 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 511.84.01081 Boehringer Ingelheim Investigational Site, Bingham Farms, Michigan
  - 511.84.01147 Boehringer Ingelheim Investigational Site, Bingham Farms, Michigan
  - 511.84.01041 Boehringer Ingelheim Investigational Site, Detroit, Michigan
  - 511.84.01131 Boehringer Ingelheim Investigational Site, Chaska, Minnesota
  - 511.84.01128 Boehringer Ingelheim Investigational Site, Chesterfield, Missouri
  - 511.84.01051 Boehringer Ingelheim Investigational Site, Kansas City, Missouri
  - 511.84.01034 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 511.84.01042 Boehringer Ingelheim Investigational Site, Billings, Montana
  - 511.84.01156 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 511.84.01148 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 511.84.01206 Boehringer Ingelheim Investigational Site, Moorestown, New Jersey
  - 511.84.01010 Boehringer Ingelheim Investigational Site, New Brunswick, New Jersey
  - 511.84.01045 Boehringer Ingelheim Investigational Site, Albequerque, New Mexico
  - 511.84.01050 Boehringer Ingelheim Investigational Site, Endwell, New York
  - 511.84.01066 Boehringer Ingelheim Investigational Site, Poughkeepsie, New York
  - 511.84.01187 Boehringer Ingelheim Investigational Site, Purchase, New York
  - 511.84.01038 Boehringer Ingelheim Investigational Site, Rochester, New York
  - 511.84.01059 Boehringer Ingelheim Investigational Site, The Bronx, New York
  - 511.84.01178 Boehringer Ingelheim Investigational Site, Chapel Hill, North Carolina
  - 511.84.01121 Boehringer Ingelheim Investigational Site, New Bern, North Carolina
  - 511.84.01119 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 511.84.01072 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 511.84.01106 Boehringer Ingelheim Investigational Site, Beachwood, Ohio
  - 511.84.01008 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.84.01062 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.84.01089 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.84.01197 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.84.01201 Boehringer Ingelheim Investigational Site, Cincinnati, Ohio
  - 511.84.01009 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.84.01014 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.84.01152 Boehringer Ingelheim Investigational Site, Cleveland, Ohio
  - 511.84.01136 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.84.01149 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.84.01151 Boehringer Ingelheim Investigational Site, Columbus, Ohio
  - 511.84.01150 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 511.84.01190 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 511.84.01112 Planned Parenthood of Arkansas & Estrn Oklahoma, Inc, Tulsa, Oklahoma
  - 511.84.01185 Boehringer Ingelheim Investigational Site, Tulsa, Oklahoma
  - 511.84.01019 Boehringer Ingelheim Investigational Site, Eugene, Oregon
  - 511.84.01134 Boehringer Ingelheim Investigational Site, Medfod, Oregon
  - 511.84.01103 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 511.84.01088 Boehringer Ingelheim Investigational Site, Jenkintown, Pennsylvania
  - 511.84.01067 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 511.84.01153 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 511.84.01145 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 511.84.01054 Boehringer Ingelheim Investigational Site, West Reading, Pennsylvania
  - 511.84.01021 Boehringer Ingelheim Investigational Site, Wilkes-Barre, Pennsylvania
  - 511.84.01060 Boehringer Ingelheim Investigational Site, Warwick, Rhode Island
  - 511.84.01063 Boehringer Ingelheim Investigational Site, Anderson, South Carolina
  - 511.84.01124 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 511.84.01123 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 511.84.01109 Boehringer Ingelheim Investigational Site, Mt. Pleasant, South Carolina
  - 511.84.01174 Boehringer Ingelheim Investigational Site, Germantown, Tennessee
  - 511.84.01163 Boehringer Ingelheim Investigational Site, Knoxville, Tennessee
  - 511.84.01026 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.84.01100 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 511.84.01078 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 511.84.01052 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 511.84.01027 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 511.84.01140 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 511.84.01084 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 511.84.01057 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.84.01082 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.84.01198 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 511.84.01036 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.84.01071 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.84.01083 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.84.01086 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 511.84.01098 Boehringer Ingelheim Investigational Site, Waco, Texas
  - 511.84.01015 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah
  - 511.84.01180 Boehringer Ingelheim Investigational Site, Sandy City, Utah
  - 511.84.01028 Boehringer Ingelheim Investigational Site, Burlington, Vermont
  - 511.84.01031 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 511.84.01035 Boehringer Ingelheim Investigational Site, Charlottesville, Virginia
  - 511.84.01107 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.84.01125 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 511.84.01076 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.84.01097 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.84.01196 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 511.84.01093 Boehringer Ingelheim Investigational Site, Bellevue, Washington
  - 511.84.01141 Boehringer Ingelheim Investigational Site, Renton, Washington
  - 511.84.01012 Boehringer Ingelheim Investigational Site, Seattle, Washington
  - 511.84.01116 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 511.84.01105 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 511.84.01177 Boehringer Ingelheim Investigational Site, Middleton, Wisconsin
- Canada (23):
  - 511.84.02007 Boehringer Ingelheim Investigational Site, Calgary, Alberta
  - 511.84.02014 Boehringer Ingelheim Investigational Site, Coquitlam, British Columbia
  - 511.84.02002 Boehringer Ingelheim Investigational Site, North Vancouver, British Columbia
  - 511.84.02021 Boehringer Ingelheim Investigational Site, Surrey, British Columbia
  - 511.84.02013 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 511.84.02015 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 511.84.02023 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 511.84.02017 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 511.84.02010 Boehringer Ingelheim Investigational Site, Woodstock, New Brunswick
  - 511.84.02012 Boehringer Ingelheim Investigational Site, Mount Pearl, Newfoundland and Labrador
  - 511.84.02006 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 511.84.02003 Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - 511.84.02018 Boehringer Ingelheim Investigational Site, Barrie, Ontario
  - 511.84.02009 Boehringer Ingelheim Investigational Site, Burlington, Ontario
  - 511.84.02022 Boehringer Ingelheim Investigational Site, London, Ontario
  - 511.84.02024 Boehringer Ingelheim Investigational Site, London, Ontario
  - 511.84.02001 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.84.02008 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 511.84.02011 Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - 511.84.02019 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 511.84.02020 Boehringer Ingelheim Investigational Site, Québec, Quebec
  - 511.84.02005 Boehringer Ingelheim Investigational Site, Sherbrooke, Quebec
  - 511.84.02004 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Jayne C, Simon JA, Taylor LV, Kimura T, Lesko LM; SUNFLOWER study investigators. Open-label extension study of flibanserin in women with hypoactive sexual desire disorder. J Sex Med. 2012 Dec;9(12):3180-8. doi: 10.1111/j.1743-6109.2012.02942.x. Epub 2012 Oct 11. PMID 23057791

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Flibanserin
Started | 1723
Completed | 667
Not Completed | 1056

BASELINE CHARACTERISTICS:
Arm/Group | Flibanserin
Number analyzed (Participants) | 1723
Age, Customized [Number; unit: participants]
  18-29 years | 266
  30-39 years | 749
  40-49 years | 672
  50 years and older | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1723
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 1492
  White Hispanic | 85
  Black | 119
  Black Hispanic | 6
  Asian | 21

OUTCOME MEASURES:

1. Primary Outcome: The Frequency of Adverse Events (Side Effects).
Description: This is a 52-week, open label trial assessing safety/tolerability of flibanserin in women with Hypoactive Sexual Desire Disorder
Time Frame: 52 weeks
Measure: Number; unit: participants with any adverse event
Arm/Group | Flibanserin
Number analyzed (Participants) | 1723
participants with any adverse event | 1272

ADVERSE EVENTS:
Arm/Group | Flibanserin
Serious Adverse Events (participants affected / at risk) | 15/1723
Other Adverse Events (participants affected / at risk) | 995/1723
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin (N=1723)
Abdominal abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Malignant melonoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flibanserin (N=1723)
Somnolence (Nervous system disorders) | 275 (315)
Fatigue (Nervous system disorders) | 131 (142)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 123 (139)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 124 (135)
Dizziness (Nervous system disorders) | 120 (152)
Headache (Nervous system disorders) | 113 (156)
Nausea (Gastrointestinal disorders) | 109 (132)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No